CLINICAL TRIAL: NCT04612595
Title: The Association Between Serum Urea Nitrogen to Creatinine Ratio and the Survival in Patients With DKD
Brief Title: The Association Between sUCR and the Survival in Patients With DKD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: WJWang002
Record Dates: First submitted 2020-06-15; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-04

CONDITIONS: Diabetic Kidney Disease
Keywords: serum urea nitrogen to creatinine ratio; diabetic kidney disease; survival
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group A: Group A are males with CKD stage 1-2.
  Interventions: Other: serum urea nitrogen to creatinine ratio
- Group B: Group B are males with CKD stage 3-4.
  Interventions: Other: serum urea nitrogen to creatinine ratio
- Group C: Group C are females with CKD stage 1-2.
  Interventions: Other: serum urea nitrogen to creatinine ratio
- Group D: Group D are females with CKD stage 3-4.
  Interventions: Other: serum urea nitrogen to creatinine ratio

INTERVENTIONS:
Other: serum urea nitrogen to creatinine ratio — According to sex and CKD stage , patients are divided into four groups,then evaluate whether the different mean sUCR and ΔsUCR can influent the survival of DKD patients.

SUMMARY:
Research Objective: To evaluate the prognostic value of serum urea nitrogen to creatinine ratio (sUCR) in the progression of DKD.

Research Design: This study was designed as a multicenter, retrospective cohort study. According to sex and CKD stage , patients are divided into four groups,then evaluate the prognostic value of mean sUCR and ΔsUCR (fluctuation of sUCR over time, meaning monthly rate of change) in the progression of DKD.

DETAILED DESCRIPTION:
Object and source: Patients diagnosed with DKD who meet the inclusion criteria are enrolled into the study.

Observation index: At baseline and every medical visit, therapeutic relevant information was collected. Data mainly include demographic characteristics(age, gender, place of residence, marriage, education degree), lifestyles(smoking, drinking, exercise), clinical characteristics(body mass index, blood pressure, duration , history of CVD, complications, nutrition situation), laboratory indexes (serum creatinine, blood urea nitrogen, glycosylated hemoglobin, urinary albumin to creatinine ratio, 24-hour urinary albumin, 24-hour urine urea nitrogen, etc.).

Quality assurance plan: The present study should be performed according to the principles of the Declaration of Helsinki and has been approved by the Ethics Committee of Guangdong Provincial People's Hospital.

Plan for missing data: When the participants drop out, the researcher should contact the participants by phone, email, text message, letter etc. and ask the reason, making record as full as possible.

Statistical analysis plan: Data are presented as mean±SD for continuous variables and as a number(percentage) for categorical variables. According to sex and CKD stage , patients are divided into four groups,then evaluate the prognostic value of mean sUCR and ΔsUCR (fluctuation of sUCR over time, meaning monthly rate of change) in the progression of DKD. The relationship between baseline characteristics among the four groups was compared by using one-way analysis of variance test, Kruskal-Wallis test or Chi-squared test where appropriate. Survival rates are estimated using Kaplan-Meier analysis, and the significance of differences was analyzed using the log-rank test. Cox proportional hazard regression analysis is used to assess the association between the clinical outcomes and mean sUCR and ΔsUCR. In multivariate analysis, we enter variables using a P value of <0.10 as the selection criterion or considered clinically significant. Hazard ratios (HRs) are presented with 95% CIs. All statistical analysis was performed with the use of SPSS (version 19.0, SPSS, Chicago, USA) and Prism 7.0 (GraphPad Software, San Diego, CA, USA). A two-tailed P value <0.05 was considered to be statistically significant.

ELIGIBILITY:
Inclusion criteria:

* Patients were diagnosed with DKD, and CKD stages 1-4.

  * Patients' age was between 18-70 years old. ③Clinical datum were complete.

Exclusion criteria:

①Patients were combined with other type of kidney disease; ②Pregnancy women; ③Infection; ④Severe liver disease; ⑤ malignant tumor;⑥Acute heart failure; ⑦Acute cardiovascular and cerebrovascular diseases ⑧gastrointestinal hemorrhage.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: DKD was defined as those diagnosed by pathological biopsy, or those with eGFR <60 ml/min per 1.73 m2, or presence of clinically detectable albuminuria over 3 months which is caused by diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
all-cause death | 10 years
  according to the criteria of death
a composite of end-stage kidney disease | 10 years
  dialysis, transplantation, or a sustained estimated GFR of <15 ml per minute per 1.73 m2
increasing by 50% of the serum creatinine level from baseline | 10 years
  increasing by 50% of the serum creatinine level from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Wenjian Wang, PhD, Study Chair — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang L, Gao P, Zhang M, Huang Z, Zhang D, Deng Q, Li Y, Zhao Z, Qin X, Jin D, Zhou M, Tang X, Hu Y, Wang L. Prevalence and Ethnic Pattern of Diabetes and Prediabetes in China in 2013. JAMA. 2017 Jun 27;317(24):2515-2523. doi: 10.1001/jama.2017.7596. PMID 28655017
- [Background] Zhang L, Long J, Jiang W, Shi Y, He X, Zhou Z, Li Y, Yeung RO, Wang J, Matsushita K, Coresh J, Zhao MH, Wang H. Trends in Chronic Kidney Disease in China. N Engl J Med. 2016 Sep 1;375(9):905-6. doi: 10.1056/NEJMc1602469. No abstract available. PMID 27579659
- [Background] Kitada M, Ogura Y, Monno I, Koya D. A Low-Protein Diet for Diabetic Kidney Disease: Its Effect and Molecular Mechanism, an Approach from Animal Studies. Nutrients. 2018 Apr 27;10(5):544. doi: 10.3390/nu10050544. PMID 29702558
- [Background] Metzger M, Yuan WL, Haymann JP, Flamant M, Houillier P, Thervet E, Boffa JJ, Vrtovsnik F, Froissart M, Bankir L, Fouque D, Stengel B. Association of a Low-Protein Diet With Slower Progression of CKD. Kidney Int Rep. 2017 Aug 30;3(1):105-114. doi: 10.1016/j.ekir.2017.08.010. eCollection 2018 Jan. PMID 29340320
- [Background] Song M, Fung TT, Hu FB, Willett WC, Longo VD, Chan AT, Giovannucci EL. Association of Animal and Plant Protein Intake With All-Cause and Cause-Specific Mortality. JAMA Intern Med. 2016 Oct 1;176(10):1453-1463. doi: 10.1001/jamainternmed.2016.4182. PMID 27479196
- [Background] Bross R, Noori N, Kovesdy CP, Murali SB, Benner D, Block G, Kopple JD, Kalantar-Zadeh K. Dietary assessment of individuals with chronic kidney disease. Semin Dial. 2010 Jul-Aug;23(4):359-64. doi: 10.1111/j.1525-139X.2010.00743.x. Epub 2010 Jul 29. PMID 20673254
- [Background] Maroni BJ, Steinman TI, Mitch WE. A method for estimating nitrogen intake of patients with chronic renal failure. Kidney Int. 1985 Jan;27(1):58-65. doi: 10.1038/ki.1985.10. PMID 3981873
- [Background] Kopple JD, Coburn JW. Evaluation of chronic uremia. Importance of serum urea nitrogen, serum creatinine, and their ratio. JAMA. 1974 Jan 7;227(1):41-4. doi: 10.1001/jama.227.1.41. No abstract available. PMID 4859625
- [Background] Inaguma D, Koide S, Ito E, Takahashi K, Hayashi H, Hasegawa M, Yuzawa Y; AICOPP group. Ratio of blood urea nitrogen to serum creatinine at initiation of dialysis is associated with mortality: a multicenter prospective cohort study. Clin Exp Nephrol. 2018 Apr;22(2):353-364. doi: 10.1007/s10157-017-1458-x. Epub 2017 Aug 1. PMID 28766029
- [Background] American Diabetes Association. 10. Microvascular Complications and Foot Care: Standards of Medical Care in Diabetes-2018. Diabetes Care. 2018 Jan;41(Suppl 1):S105-S118. doi: 10.2337/dc18-S010. PMID 29222381

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT04612595/Prot_SAP_000.pdf